CLINICAL TRIAL: NCT02795650
Title: Personalised Therapy for Patients With Metastatic Adenocarcinoma of the Pancreas Determined by Genetic Testing and Avatar Model Generation
Brief Title: Personalised Therapy for Metastatic ADPC Determined by Genetic Testing and Avatar Model Generation
Acronym: AVATAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario de Fuenlabrada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004860-12
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Adenocarcinoma
Keywords: Metastatic; Pancreas
MeSH Terms: conditions — Adenocarcinoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): Personalised treatment will be chosen for patients based on the results of tumor sequencing, bioinformatics and avatar model drug testing.
  Interventions: Drug: Personalised treatment
- Control (Active Comparator): Investigators are allowed to chose the best option of standard treatment for patients.
  Interventions: Drug: Treatment chosen per investigator´s judge

INTERVENTIONS:
Drug: Personalised treatment — Personalised treatments include chemotherapy, targeted therapy, immunotherapy or others based on the previous test results, chosen from a database that include more than 2000 different drugs.
  Arms: Experimental arm
Drug: Treatment chosen per investigator´s judge — Investigators are allowed to chose what they consider the best standard treatment option for their patients.
  Arms: Control

SUMMARY:
This is a multicenter, open label, randomised phase II clinical trial for patients with metastatic adenocarcinoma of the pancreas. Patients randomised to the experimental arm will undergone tumoral biopsy before starting first line of treatment and will be administered personalised therapy as second or third line.

DETAILED DESCRIPTION:
This is a multicenter, open label, randomised phase II clinical trial for patients with metastatic adenocarcinoma of the pancreas.

Patients with metastatic disease will be randomised to the experimental or control arms. Those in the experimental arm will undergone a tumoral biopsy in order to perform exome sequencing, bioinformatic report, and avatar mouse models for drug testing. This information will allow the expertise panel to elaborate a treatment recommendation as second or third lines of treatment. Patients in the control arm will receive treatment as per investigator´s judge. The main objective of the trial is to determine whether personalised treatments achieve improved 1-year overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the pancreas.
* ECOG performance status 0 or 1
* Age ≥ 18 years old.
* Willingness of male and female subjects, who are not surgically sterile or postmenopausal, to use reliable methods of birth control (oral contraceptives, intrauterine devices, or barrier methods used with a spermicide) for the duration of the study.
* One or more sites of metastasis with one of the susceptible of biopsy.
* Measurable or evaluable disease
* No prior treatment with radiotherapy, surgery, chemotherapy or investigational treatment for the metastatic disease or no more than the three cycles of first line chemotherapy. Palliative radiotherapy for bone metastasis is allowed. Adjuvant or neoadjuvant radiotherapy or chemotherapy are allowed if they finished more that 6 months ago and the patient has no remaining toxicities.
* Bone marrow function as follows, no more than 14 days prior to randomisation:

ANC > 1,500 cells/mm3 Platelets > 100,000 cells/mm3 Hemoglobin ≥9 g/dl

* Adequate liver, renal and bone marrow functions.

  * AST (SGOT), ALT (SGPT) ≤ 2.5 × ULN and ≤ 5 x ULN if liver metastases.
  * Bilirubin ≤ 1,5 x ULN
  * Albumin total ≥ 0,75 ULN
  * Creatinine ≤ 1,5 x ULN
* Ability to sign informed consent
* Patients will be allowed to be randomised just once.

Exclusion Criteria:

* Brain metastases, unless they have been previously treated and stable for 3 months at least (defined as no oedema, no need of steroids and stable disease in two CT scans separated by a minimum of 4 weeks).
* Locally advanced disease.
* Malignancies other than pancreatic cancer diagnosed within 5 years prior to randomization, except for adequately treated carcinoma in situ or basal or squamous cell skin cancer.
* Bacterial, viral or fungal active infection that require systemic treatment.
* Any contraindication for tumor biopsy.
* Past or present HIV or hepatitis B or C infection.
* Severe medical problems affecting organs or psychiatric illnesses that could interfere with the safety of the patient in the trial.
* Pregnancy or breastfeeding women.
* Patient will need to be informed and agree to undergo tumoral biopsy in the experimental arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
1-year overall survival | 1-year overall survival
  Efficacy. 1-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- Spain (5):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de la Paz, Madrid
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huebner A, Black JRM, Sarno F, Pazo R, Juez I, Medina L, Garcia-Carbonero R, Guillen C, Feliu J, Alonso C, Arenillas C, Moreno-Cardenas AB, Verdaguer H, Macarulla T, Hidalgo M, McGranahan N, Toledo RA. ACT-Discover: identifying karyotype heterogeneity in pancreatic cancer evolution using ctDNA. Genome Med. 2023 Apr 20;15(1):27. doi: 10.1186/s13073-023-01171-w. PMID 37081523